CLINICAL TRIAL: NCT02354027
Title: Drug Interaction Study of Henagliflozin and Metformin in Healthy Subjects
Brief Title: The Drug-drug Interaction of SHR3824 and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-105
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824 metformin drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR3824 25mg/metformin 1000mg (Experimental): Two 500-mg tablets of metformin on Day 1 followed by 25 mg of SHR3824 once daily on Days 4 through 8 followed by two 500-mg tablets of metformin and 25 mg of SHR3824 on Day 8.
  Interventions: Drug: SHR3824 metformin

INTERVENTIONS:
Drug: SHR3824 metformin — Two 500-mg tablets of metformin on Day 1 followed by 25 mg of SHR3824 once daily on Days 4 through 8 followed by two 500-mg tablets of metformin and 25 mg of SHR3824 on Day 8.
  Drug: SHR3824 + Metformin
  Other Names: Henagliflozin metformin

SUMMARY:
The purpose of the study is to investigate the potential interaction between multiple oral doses of SHR3824 and a single oral dose of metformin in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center study of SHR3824 and metformin in healthy adult volunteers. SHR3824(a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus (T2DM) and metformin is an approved treatment for patients with T2DM. SHR3824 will be administered orally (by mouth) as 25 mg on Days 4, 5, 6, 7, and 8 and metformin will be administered orally as two 500mg tablets on Days 1 and 8. Both SHR3824 and metformin tablets will be taken with 8 ounces (240 mL) of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 24 kg/m2.

Exclusion Criteria:

* History of diabetes
* History of heart failure or renal insufficiency
* Urinary tract infections, or vulvovaginal mycotic infections
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SHR3824 or metformin or any of the excipients of the formulation of SHR3824 or metformin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR3824. | At protocol-specified times up to Day 9.
  Cmax (a measure of the body's exposure to SHR3824) will be compared before and after administration of a single dose of metformin.
The area under the plasma concentration-time curve (AUC) of SHR3824. | At protocol-specified times up to Day 9.
  AUC (a measure of the body's exposure to SHR3824) will be compared before and after administration of a single dose of metformin.
The maximum plasma concentration (Cmax) of metformin. | At protocol-specified times up to Day 9.
  Cmax (a measure of the body's exposure to metformin) will be compared. before and after administration of multiple doses of SHR3824
The area under the plasma concentration-time curve (AUC) of metformin | At protocol-specified times up to Day 9.
  AUC (a measure of the body's exposure to metformin) will be compared before and after administration of multiple doses of SHR3824.

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability. | Up tp day 9.